CLINICAL TRIAL: NCT00154531
Title: Identification of Biomarkers Associated With Human Hepatocellular Carcinoma by Surface-Enhanced Laser Desorption/Ionization (SELDI)
Brief Title: Identification of Biomarkers Associated With Human Hepatocellular Carcinoma by SELDI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9261701418
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-12-20 (Estimated); Status verified 2003-12

CONDITIONS: Hepatocellular Carcinoma; Hepatitis B; Hepatitis C
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis B; Hepatitis C

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Hepatocellular carcinoma (HCC) has been the leading cause of cancer death in Taiwan. Though Alpha-fetoprotein (AFP) and des-γ-carboxy prothrombin(DCP) are used as the tumor markers for diagnosis of HCCs. Thus, these two markers are not good enough for the early detection of small HCCs. To improve the survival, further investigations of the early diagnostic markers are still needed.

SELDI is a proteomic profiling techniques in biomarker discovery. Its approach has been successfully used to identify biomarkers of various cancers, such as prostate cancer, bladder cancer, ovarian cancer, lung cancer, colon cancer, breast cancer and pancreatic cancer.

In this current project we will apply the SELDI technique to identify the HCC biomarkers. Sera samples from the HCC patients and relevant controls will be collected. We hope that we can find the new HCC biomarkers. If biomarkers of HCC are identified, this can be used to clinical application for the possible early detection of HCCs.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) has been the leading cause of cancer death in Taiwan. Above 6000-8000 people died of this cancer every year in Taiwan. Though regular sonographic examination can early detect small HCC and there are many therapeutic modalities for HCC, the therapeutic results remains unsatisfactory. Though Alpha-fetoprotein (AFP) and des-γ-carboxy prothrombin(DCP) are used as the tumor markers for diagnosis of HCCs, AFP is normal in around one third of small(<3cm) HCC patients. Elevated DCP activities were present in 44%-47.6% with HCCs less than 3cm. Thus, these two markers are not good enough for the early detection of small HCCs. To improve the survival, further investigations of the early diagnostic markers are still needed.

The global analysis of cellular proteins has recently been termed proteomics and is a key area if research that is developing in the postgenomic ear. With respect to cancer, proteomics has the potential to identify novel targets for therapy or markers for diagnosis. The proteomic profiling techniques in biomarker discovery include (1) 2-D PAGE / MALDI-MS (two-dimensional gel electrophoresis, polyacrylamide gel electrophoresis) / matrix assisted laser desorption / ionization-mass spectrometry), (2) LC/MS/MS (liquid chromatography/MS/MS), (3) SELDI-TOF (surface-enhanced laser desorption ionization time-of-flight). These techniques have their own advantages and shortcomings.

SELDI is a recently descried modification of MALDI-TOP in which small amounts of protein are directly applied to a biochip coated with specific chemical matrices (hydrophobic, cationic, anionic, normal phase, and so forth) or biochemical molecules such as DNA oligonucleotides or purified proteins. The bound proteins retained after washing are analyzed by mass spectrometry to obtain the protein fingerprint of the sample. The detected proteins are displayed as a series of peaks.

SELDI-TOF MS can offer high-throughput protein profiles. Blood, urine, body fluid, or tissue specimen are taken from the patients and then are applied onto different ProteinChip Arrays. The differences in the protein expression profiles of two or more distinct samples are thus obtained. SELDI approach has been successfully used to identify biomarkers of various cancers, such as prostate cancer, bladder cancer, ovarian cancer, lung cancer, colon cancer, breast cancer and pancreatic cancer.

In this current project we will apply the SELDI technique to identify the HCC biomarkers. Sera samples from the HCC patients and relevant controls will be collected. The samples will then be applied to SELDI analysis. We hope that we can find the new HCC biomarkers. If biomarkers of HCC are identified, this can be used to clinical application for the possible early detection of HCCs.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hepatocellular carcinoma
* Clinical diagnosis of hepatitis B
* Clinical diagnosis of hepatitis C

Exclusion Criteria:

* N/A

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 230
Dates: Start 2004-08; Study Completion 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Chuan Sheu, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan